CLINICAL TRIAL: NCT02549456
Title: Natural Orifice Transluminal Endoscopic Surgery for Colorectal Cancer
Acronym: NOTES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Collaborators: Universidade da Coruña (Other)
Responsible Party: Principal Investigator, Islam Hany Metwally, Assistant lecturer of surgical oncology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD/148
Record Dates: First submitted 2015-08-29; First posted 2015-09-15 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Cancer
Keywords: natural orifice surgery; natural orifice specimen extraction; taTME
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Natural orifice specimen extraction (Experimental): Conventional laparoscopic resection of colorectal cancer with natural orifice specimen extraction
  Interventions: Procedure: natural orifice specimen extraction
- Laparoendoscopic resection (Experimental): Laparoscopic assisted transanal endoscopic resection of rectal cancer
  Interventions: Procedure: Laparoendoscopic resection

INTERVENTIONS:
Procedure: natural orifice specimen extraction — Conventional laparoscopic resection of colorectal cancer is done then specimen is extracted through natural orifice (anal or vaginal orifice).
  Arms: Natural orifice specimen extraction
Procedure: Laparoendoscopic resection — Endoscopic phase: Transanal platform is inserted into the rectum, and pneumorectum is established. The lumen is occluded below the level of the tumor. The avascular ''oncologic'' presacral plane is entered posteriorly, and dissection proceeds cephalad in the total mesorectal excision planes. Next, the abdominal cavity is entered at the peritoneal reﬂection. The superior rectal artery is divided. The rectal stump then is reﬂected into the abdominal cavity, and retrograde dissection is performed until the procedure is limited by instrument length.
  Laparoscopic phase: Colon mobilization, lymph node dissection, and mesenteric excision are performed laparoscopically. Mobilization of the splenic ﬂexure is done if needed.
  Arms: Laparoendoscopic resection

SUMMARY:
The purpose of this study is to assess different hybrid natural orifice transluminal endoscopic surgery techniques in management of colorectal cancer as regard: feasibility of the technique, short term oncologic outcome and functional outcome.

DETAILED DESCRIPTION:
Intervention will be done by conventional laparoscopy and transanal endoscopy (TEO or Gelpoint platform), patients are divided into two arms to compare different natural orifice techniques in resection of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Medically fit patient.
2. Non metastatic pathologically proven sigmoid colon cancer.
3. Non metastatic pathologically proven rectal cancer.
4. Patient continent for stool.

Exclusion Criteria:

1. Patients with American Society of Anesthesiologist (ASA) score 4 and 5.
2. Patients with cardiac or chest problems that cannot withstand insufflation.
3. Unresectable tumors (defined as those who cannot be resected without a high likelihood of leaving microscopic or gross residual disease at the local site because of tumor adherence or fixation).
4. Obstructed or perforated cancer.
5. Patients with metastatic colorectal cancer.
6. Incontinent patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 24 hour
  Rate of conversion to classic laparoscopy or to open laparotomy.
operative time | 24 hour
  time taken from starting operation till patient wake up
Operative blood loss | 24 hour
  measured in milliliter
Wound complications | two week
  infection-dehiscence
Major intraoperative complications | 24 hour
  bleeding -organ injury
Major postoperative complications | two weeks
  leak-bleeding

SECONDARY OUTCOMES:
Adequacy of lymphadenectomy | one month
  Number of lymph nodes retrieved
Grading of quality and completeness of mesorectal excision | one month
  It is a composite outcome where result will appear as either complete, near complete or incomplete. Criteria in (shape, coning, presence of defects and circumferential safety margin) will be integrated to categorize it.
Longitudinal safety margin | one month
  either free or infiltrated with tumor by histopathology examination.
short term oncologic outcome | 6 months - one year
  incidence of local and distant outcomes and disease free survival
Functional outcome | 3 months
  assessing fecal incontinence using Kirwan's grading score

CONTACTS AND LOCATIONS:
Overall Officials: Jose F Noguira, MD, Study Director — Head of general and digestive surgery department, CHUAC, universidade da Coruna; Sherif Z Kotb, MD, Study Chair — Professor of surgical oncology, Oncology center Mansoura University
Locations (1):
- Oncology center Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt